CLINICAL TRIAL: NCT01699789
Title: CPIC is a Community Partnered Participatory Research (CPPR) Project of Community and Academic Partners Working Together to Learn the Best Way to Reduce Depression in Our Communities.
Brief Title: Community Partners in Care is a Research Project Funded by the National Institutes of Health
Acronym: CPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Robert Wood Johnson Foundation (Other); National Library of Medicine (NLM) (NIH); Patient-Centered Outcomes Research Institute (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CPIC-2012-KW; R01MH078853 (NIH); P30MH082760 (NIH); P30MH068639 (NIH); PPRN-1501-26518 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute); R01MD007721 (NIH); G08LM011058 (NIH); UL1TR000124 (NIH); 64244 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Depression; Information Dissemination; Social Determinants of Health
Keywords: Community Partnered Participatory Research; Community Engagement; Implementation; Community Based Participatory Research; Quality Improvement; Evidence Based Practice; Patient Centered Outcomes Research
MeSH Terms: conditions — Depression | interventions — Health Resources

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resources for Services (Active Comparator): The Resources for Services condition offers time-limited technical assistance to individual agencies, coupled with outreach from a community engagement specialty, to participate in structured reviews of components of the Quality Improvement Program Intervention as implemented by the Resources for Services Expert Team.
  Interventions: Other: Quality Improvement Program; Behavioral: Resources for Services Expert Team
- Community Engagement and Planning (Experimental): The Community Engagement and Planning arm supported 4 months of planning for the Community Engagement and Planning Council consisting representatives of all assigned programs in biweekly 2 hour meetings to fit trainings in the Quality Improvement Program to the community and develop strategies across programs to collaborate as a network. The CEP Council developed a written plan for training and monitoring and supported implementation of the training plan. CEP sites were provided with enrolled client lists.
  Interventions: Other: Quality Improvement Program; Behavioral: Community Engagement and Planning Council

INTERVENTIONS:
Other: Quality Improvement Program — The quality improvement program is an evidence-based toolkit from prior studies (see Names above) that supported team leadership, case and care management, medication management, and Cognitive Behavioral Therapy for Depression. The Case management manual supported depression screening and monitoring/tracking of outcomes; patient education and activation, care coordination, and behavioral activation and problem solving. The toolkit includes education on depression and a community health worker manual.
  Other Names: Partners in Care; We Care; IMPACT; Mental Health Infrastructure and Training Project
Behavioral: Resources for Services Expert Team — The expert team consisted for RS consisted of 3 psychiatrists, a psychologist expert in Cognitive Behavioral Therapy, a nurse care manager, a community engagement specialist, a quality improvement expert, and staff support. They team offered 12 web-based seminars to each community on components of collaborative care as well as site visits to primary care clinics on clinical assessment and medication management.
  Other Names: Quality Improvement Team
  Arms: Resources for Services
Behavioral: Community Engagement and Planning Council — The CEP Council was supported by a workbook developed by the overall CPIC Council that provided principles, approach, agendas, and resources for the multi-sector planning meetings. The CEP Councils met twice a month for 4-6 months to develop their plan and met monthly during implementation of trainings. The study Council supported CEP meetings. Community leaders co-led trainings with study experts to help assure sustainability. Each CEP council had $15K to defray costs of venues, materials, and consultations, while the study provided that for RS.
  Other Names: Quality Improvement Team
  Arms: Community Engagement and Planning

SUMMARY:
CPIC is a community initiative and research study funded by the NIH. CPIC was developed and is being run by community and academic partners in Los Angeles underserved communities of color. CPIC compares two ways of supporting diverse health and social programs in under-resourced communities to improve their services to depressed clients. One approach is time-limited expert technical assistance coupled with culturally-competent community outreach to individual programs, on how to use quality improvement toolkits for depression that have already been proven to be effective or helpful in primary care settings, but adapted for this study for use in diverse community-based programs in underserved communities. The other approach brings different types of agencies and members in a community together in a 4 to 6-month planning process, to fit the same depression quality improvement programs to the needs and strengths of the community and to develop a network of programs serving the community to support clients with depression together. The study is designed to determine the added value of community engagement and planning over and above what might be offered through a community-oriented, disease management company. Both intervention models are based on the same quality improvement toolkits that support team leadership, care management, Cognitive Behavioral Therapy, medication management, and patient education and activation. Investigators hypothesized that the community engagement approach would increase agency and clinician participation in evidence-based trainings and improve client mental health-related quality of life. In addition, during the design phase, community participants prioritized adding as outcomes indicators of social determinants of mental health, including physical functioning, risk factors for homelessness and employment. Investigators hypothesized by activating community agencies that can address health and social services needs to engage depressed clients, these outcomes would also be improved more in the collaboration condition. Investigators also hypothesized that the collaboration approach would increase use of services.

DETAILED DESCRIPTION:
Underserved communities of color in low income, largely ethnic-minority neighborhoods face an excessive burden of illness from depression due to higher prevalence of depression and lower access to quality care. Evidence-based quality improvement (QI) programs for depression in primary care settings-where many low-income and minority patients receive their only mental health care-can enhance quality of depression care and improve health outcomes. These programs are under-utilized in community-based health care settings, and have not been adapted for use across diverse agencies (social service, faith based, primary and specialty care) that could partner to support disease management for depression. Partners in Care (PIC)and WE Care are interventions designed to improve access to evidence-based depression treatments (medication management or psychotherapy) for primary care patients and, in WE Care, social service clients. PIC evaluated a services delivery intervention while WE Care was an effectiveness trial with study-provided treatments. Both studies promoted use of the same evidence-based treatments. Both PIC and WE Care programs improved use of evidence-based treatments for depression and health outcomes for African Americans and Latinos. The PIC interventions reduced health outcome disparities evident in usual care in the first follow-up year and at five-year follow-up. While these findings offer hope to underserved communities, such communities have poor resources to support implementation of these programs, and may have historical distrust in research and health care settings. There is no evidence-based approach to support agency networks in underserved communities in implementing QI programs for depression. To address this information gap, investigators created Community Partners in Care (CPIC), a group-level randomized, controlled trial, with randomization at the level of an agency site or "unit." The trial is being fielded in two underserved communities, Hollywood and South Los Angeles, and conducted through a community- participatory, partnered research (CPPR) approach.

The specific aims of the study are:

1. To engage two underserved communities in improving safety-net care for depression.
2. To examine the effects of a community-engagement approach to implementing evidence-based depression quality improvement toolkits (PIC/WE Care) through a community collaborative network across services sectors, compared to technical assistance to individual programs from the same services sectors coupled with culturally-competent outreach to implement the same toolkits. The outcomes are: a) client access to care, quality of care and health outcomes, with the primary outcome being mental-health related quality of life and additional outcomes reflecting social determinants of mental health of interest to the community (physical health, homelessness risk factors, employment); b) services utilization and costs; c) agency adoption of PIC/WE Care; d) and provider attitudes, knowledge and practice.
3. To describe the process of implementation of the community engagement intervention.

CPIC was awarded funds from the Patient Centered Outcomes Research Institute (PCORI) in 2013 to accomplish the following 3 aims:

1. To compare the long-term (3-year) effectiveness of community engagement and planning versus agency technical assistance to implement depression QI and improve depressed clients' health status and risk for homelessness
2. To determine how depressed clients in under-resourced communities prioritize diverse health and social outcomes and identify their preferences for services to address priority outcomes
3. To identify capacities of providers to respond to depressed clients' priorities and to generate recommendations for building capacity to better address clients'priorities.

We hypothesize that community engagement and planning will be more effective than technical assistance in improving 3-year outcomes and that clients will prioritize quality of life. We expect to find gaps in provider capacities to address client priorities that network strategies could address.

Our primary outcome for the long-term follow-up is mental health related quality of life and secondary outcomes are use of healthcare and community services for depression and physical functioning and homeless risk factors.

In 2014, CPIC was awarded funds from the National Institute on Minority Health and Health Disparities (NIMHD) to use existing quantitative CPIC data and collect new qualitative data to describe pathways to reducing disparities. The funding allows us to longitudinally track the implementation of the CEP model in a new county-wide initiative to develop community networks to promote healthy neighborhoods. The aims under this additional funding are:

1. To determine pathways to reducing mental health and social disparities by conducting community-academic partnered analyses of CPIC data by 1) examining intervention effects for disparity subgroups (African Americans, Latinos, gender groups, insurance and housing status groups); 2) identifying predictors and mediators of barriers to access/services and client outcomes; 3) analyzing intervention effects on provider workforce diversity; and 4) generating explanatory models for intervention effects and their sustainability by interviewing CPIC administrators and providers, as well as prior and current clients.
2. To explore the generalizability and replicability of the CPIC partnered model and, more broadly, to inform the process of incorporating science into policy by conducting a longitudinal case study of the CEP model implementation in a county-wide "neighborhood health" initiative in Los Angeles to reduce mental health and social disparities.

As a result of this study, we will be able to explain how community-engaged and participatory models of intervention implementation can reduce health and social disparities and ultimately achieve public health impact. Study findings will be disseminated widely using traditional academic, community-valued, and policy-relevant dissemination channels.

ELIGIBILITY:
Inclusion Criteria:

Administrators

* Age 18 and above
* Work or volunteer for an enrolled program in the study and be designated as a liaison by the program

Providers

* Age 18 and above
* Have direct contact with patients/clients

Clients

* Age 18 and above
* Score 10 or greater on modified Patient Health Questionnaire (PHQ-8)

Exclusion Criteria: grossly disorganized by screener staff assessment Not providing personal contact information

Administrators - Under age 18

Providers

- Under age 18

Clients

* Under age 18
* Gross cognitive disorganization by screener staff assessment
* Providing no contact information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2009-01; Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth B Wells, M.D., M.P.H, Principal Investigator — RAND Corporation, UCLA Semel Institute; Bowen Chung, MD, MSHS, Principal Investigator — Harbor-UCLA Medical Center, UCLA Semel Institute; Jeanne Miranda, PhD, Principal Investigator — UCLA Semel Institute
Locations (1):
- Krystal M Griffith, Gardena, California, United States

REFERENCES:
- [Background] Chung B, Jones L, Dixon EL, Miranda J, Wells K; Community Partners in Care Steering Council. Using a community partnered participatory research approach to implement a randomized controlled trial: planning community partners in care. J Health Care Poor Underserved. 2010 Aug;21(3):780-95. doi: 10.1353/hpu.0.0345. PMID 20693725
- [Background] Khodyakov D, Mendel P, Dixon E, Jones A, Masongsong Z, Wells K. Community Partners in Care: Leveraging Community Diversity to Improve Depression Care for Underserved Populations. Int J Divers Organ Communities Nations. 2009;9(2):167-182. PMID 21528111
- [Background] Dixon EL, Flaskerud JH. Community tailored responses to depression care. Issues Ment Health Nurs. 2010 Sep;31(9):611-3. doi: 10.3109/01612841003675303. No abstract available. PMID 20701424
- [Background] Mango J, Cabiling E, Jones L, Lucas-Wright A, Williams P, Wells K, Pulido E, Meldrum M, Ramos A, Chung B. Community Partners in Care (CPIC): Video Summary of Rationale, Study Approach / Implementation, and Client 6-month Outcomes. CES4healthinfo. 2014 Feb 25;2014:87LWR5H2. PMID 25364622
- [Background] Khodyakov D, Pulido E, Ramos A, Dixon E. Community-partnered research conference model: the experience of Community Partners in Care study. Prog Community Health Partnersh. 2014 Spring;8(1):83-97. doi: 10.1353/cpr.2014.0008. PMID 24859106
- [Background] Mendel P, Ngo VK, Dixon E, Stockdale S, Jones F, Chung B, Jones A, Masongsong Z, Khodyakov D. Partnered evaluation of a community engagement intervention: use of a kickoff conference in a randomized trial for depression care improvement in underserved communities. Ethn Dis. 2011 Summer;21(3 Suppl 1):S1-78-88. PMID 22352084
- [Background] Belin TR, Jones A, Tang L, Chung B, Stockdale SE, Jones F, Wright A, Sherbourne CD, Perlman J, Pulido E, Ong MK, Gilmore J, Miranda J, Dixon E, Jones L, Wells KB. Maintaining Internal Validity in Community Partnered Participatory Research: Experience from the Community Partners in Care Study. Ethn Dis. 2018 Sep 6;28(Suppl 2):357-364. doi: 10.18865/ed.28.S2.357. eCollection 2018. PMID 30202188
- [Background] Mendel P, O'Hora J, Zhang L, Stockdale S, Dixon EL, Gilmore J, Jones F, Jones A, Williams P, Sharif MZ, Masongsong Z, Kadkhoda F, Pulido E, Chung B, Wells KB. Engaging Community Networks to Improve Depression Services: A Cluster-Randomized Trial of a Community Engagement and Planning Intervention. Community Ment Health J. 2021 Apr;57(3):457-469. doi: 10.1007/s10597-020-00632-5. Epub 2020 May 19. PMID 32430557
- [Background] Goodsmith N, Zhang L, Ong MK, Ngo VK, Miranda J, Hirsch S, Jones F, Wells K, Chung B. Implementation of a Community-Partnered Research Suicide-Risk Management Protocol: Case Study From Community Partners in Care. Psychiatr Serv. 2021 Mar 1;72(3):281-287. doi: 10.1176/appi.ps.202000095. Epub 2021 Jan 27. PMID 33502218
- [Result] Wells KB, Jones L, Chung B, Dixon EL, Tang L, Gilmore J, Sherbourne C, Ngo VK, Ong MK, Stockdale S, Ramos E, Belin TR, Miranda J. Community-partnered cluster-randomized comparative effectiveness trial of community engagement and planning or resources for services to address depression disparities. J Gen Intern Med. 2013 Oct;28(10):1268-78. doi: 10.1007/s11606-013-2484-3. Epub 2013 May 7. PMID 23649787
- [Result] Miranda J, Ong MK, Jones L, Chung B, Dixon EL, Tang L, Gilmore J, Sherbourne C, Ngo VK, Stockdale S, Ramos E, Belin TR, Wells KB. Community-partnered evaluation of depression services for clients of community-based agencies in under-resourced communities in Los Angeles. J Gen Intern Med. 2013 Oct;28(10):1279-87. doi: 10.1007/s11606-013-2480-7. Epub 2013 May 14. PMID 23670566
- [Result] Chung B, Ong M, Ettner SL, Jones F, Gilmore J, McCreary M, Sherbourne C, Ngo V, Koegel P, Tang L, Dixon E, Miranda J, Belin TR, Wells KB. 12-month outcomes of community engagement versus technical assistance to implement depression collaborative care: a partnered, cluster, randomized, comparative effectiveness trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S23-34. doi: 10.7326/M13-3011. PMID 25402400
- [Result] Chang ET, Wells KB, Gilmore J, Tang L, Morgan AU, Sanders S, Chung B. Comorbid depression and substance abuse among safety-net clients in Los Angeles: a community participatory study. Psychiatr Serv. 2015 Mar 1;66(3):285-94. doi: 10.1176/appi.ps.201300318. Epub 2014 Dec 1. PMID 25727117
- [Result] Chung B, Ngo VK, Ong MK, Pulido E, Jones F, Gilmore J, Stoker-Mtume N, Johnson M, Tang L, Wells KB, Sherbourne C, Miranda J. Participation in Training for Depression Care Quality Improvement: A Randomized Trial of Community Engagement or Technical Support. Psychiatr Serv. 2015 Aug 1;66(8):831-9. doi: 10.1176/appi.ps.201400099. Epub 2015 May 1. PMID 25930037
- [Result] Ngo VK, Sherbourne C, Chung B, Tang L, Wright AL, Whittington Y, Wells K, Miranda J. Community Engagement Compared With Technical Assistance to Disseminate Depression Care Among Low-Income, Minority Women: A Randomized Controlled Effectiveness Study. Am J Public Health. 2016 Oct;106(10):1833-41. doi: 10.2105/AJPH.2016.303304. Epub 2016 Aug 23. PMID 27552274
- [Result] Landry CM, Jackson AP, Tang L, Miranda J, Chung B, Jones F, Ong MK, Wells K. The Effects of Collaborative Care Training on Case Managers' Perceived Depression-Related Services Delivery. Psychiatr Serv. 2017 Feb 1;68(2):123-130. doi: 10.1176/appi.ps.201500550. Epub 2016 Sep 15. PMID 27629796
- [Result] Ong MK, Jones L, Aoki W, Belin TR, Bromley E, Chung B, Dixon E, Johnson MD, Jones F, Koegel P, Khodyakov D, Landry CM, Lizaola E, Mtume N, Ngo VK, Perlman J, Pulido E, Sauer V, Sherbourne CD, Tang L, Vidaurri E, Whittington Y, Williams P, Lucas-Wright A, Zhang L, Southard M, Miranda J, Wells K. A Community-Partnered, Participatory, Cluster-Randomized Study of Depression Care Quality Improvement: Three-Year Outcomes. Psychiatr Serv. 2017 Dec 1;68(12):1262-1270. doi: 10.1176/appi.ps.201600488. Epub 2017 Jul 17. PMID 28712349
- [Result] Mehta P, Brown A, Chung B, Jones F, Tang L, Gilmore J, Miranda J, Wells K. Community Partners in Care: 6-Month Outcomes of Two Quality Improvement Depression Care Interventions in Male Participants. Ethn Dis. 2017 Jul 20;27(3):223-232. doi: 10.18865/ed.27.3.223. eCollection 2017 Summer. PMID 28811733
- [Result] Castillo EG, Shaner R, Tang L, Chung B, Jones F, Whittington Y, Miranda J, Wells KB. Improving Depression Care for Adults With Serious Mental Illness in Underresourced Areas: Community Coalitions Versus Technical Support. Psychiatr Serv. 2018 Feb 1;69(2):195-203. doi: 10.1176/appi.ps.201600514. Epub 2017 Oct 16. PMID 29032700
- [Result] Sherbourne CD, Aoki W, Belin TR, Bromley E, Chung B, Dixon E, Gilmore JM, Johnson MD, Jones F, Koegel P, Khodyakov D, Landry CM, Lizaola E, Mtume N, Ngo VK, Ong MK, Perlman J, Pulido E, Sauer V, Tang L, Whittington Y, Vidaurri E, Williams P, Lucas-Wright A, Zhang L, Miranda J, Jones L, Wells K. Comparative Effectiveness of Two Models of Depression Services Quality Improvement in Health and Community Sectors. Psychiatr Serv. 2017 Dec 1;68(12):1315-1320. doi: 10.1176/appi.ps.201700170. Epub 2017 Nov 1. PMID 29089009
- [Result] Springgate B, Tang L, Ong M, Aoki W, Chung B, Dixon E, Johnson MD, Jones F, Landry C, Lizaola E, Mtume N, Ngo VK, Pulido E, Sherbourne C, Wright AL, Whittington Y, Williams P, Zhang L, Miranda J, Belin T, Gilmore J, Jones L, Wells KB. Comparative Effectiveness of Coalitions Versus Technical Assistance for Depression Quality Improvement in Persons with Multiple Chronic Conditions. Ethn Dis. 2018 Sep 6;28(Suppl 2):325-338. doi: 10.18865/ed.28.S2.325. eCollection 2018. PMID 30202185
- [Result] Choi KR, Sherbourne C, Tang L, Castillo E, Dixon E, Jones A, Chung B, Eisen C, Wells K. A Comparative Effectiveness Trial of Depression Collaborative Care: Subanalysis of Comorbid Anxiety. West J Nurs Res. 2019 Jul;41(7):1009-1031. doi: 10.1177/0193945918800333. Epub 2018 Sep 18. PMID 30226112
- [Result] Chung B, Ong M, Ettner SL, Jones F, Gilmore J, McCreary M, Ngo VK, Sherbourne C, Tang L, Dixon E, Koegel P, Miranda J, Wells KB. 12-Month Cost Outcomes of Community Engagement Versus Technical Assistance for Depression Quality Improvement: A Partnered, Cluster Randomized, Comparative-Effectiveness Trial. Ethn Dis. 2018 Sep 6;28(Suppl 2):349-356. doi: 10.18865/ed.28.S2.349. eCollection 2018. PMID 30202187
- [Result] Arevian AC, Jones F, Tang L, Sherbourne CD, Jones L, Miranda J; Community Partners in Care Writing Group. Depression Remission From Community Coalitions Versus Individual Program Support for Services: Findings From Community Partners in Care, Los Angeles, California, 2010-2016. Am J Public Health. 2019 Jun;109(S3):S205-S213. doi: 10.2105/AJPH.2019.305082. PMID 31242001
- [Result] Barcelo NE, Lopez A, Tang L, Aguilera Nunez MG, Jones F, Miranda J, Chung B, Arevian A, Bonds C, Izquierdo A, Dixon E, Wells K. Community Engagement and Planning versus Resources for Services for Implementing Depression Quality Improvement: Exploratory Analysis for Black and Latino Adults. Ethn Dis. 2019 Apr 18;29(2):277-286. doi: 10.18865/ed.29.2.277. eCollection 2019 Spring. PMID 31057313
- [Result] Morton I, Hurley B, Castillo EG, Tang L, Gilmore J, Jones F, Watkins K, Chung B, Wells K. Outcomes of two quality improvement implementation interventions for depression services in adults with substance use problems. Am J Drug Alcohol Abuse. 2020;46(2):251-261. doi: 10.1080/00952990.2019.1708085. Epub 2020 Jan 14. PMID 31935133
- See also: Click here for more information about this study: Community Partners in Care — http://www.communitypartnersincare.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 2010 to November 2010, the study screened 4,440 clients from 93 programs in 50 agencies. The ninety-three programs, included 17 primary care/public health, 18 mental health, 20 substance abuse, ten homeless services, and 28 social/other community services.
Groups:
- Resources for Services RS: The RS condition offers time-limited technical assistance to individual agencies, coupled with outreach from a community engagement specialty, to participate in structured reviews of components of the Quality Improvement (QI) Program Intervention as implemented by the RS Expert Team.
  QI Program: The quality improvement program is an evidence-based toolkit from prior studies that supported team leadership, case and care management, medication management, and CBT for Depression. The Case management manual supported depression screening and monitoring/tracking of outcomes; patient education and activation, care coordination, and behavioral activation and problem solving. The toolkit includes education on depression and a community health worker manual.
  RS Expert Team: The expert team for RS consisted of 3 psychiatrists, a psychologist expert in CBT, a nurse care manager, a community engagement specialist, a quality improvement expert, and staff support. T
- Community Engagement and Planning CEP: The CEP arm supported 4 months of planning for the CEP Council consisting of representatives from all assigned programs in biweekly 2 hour meetings to fit trainings in the QI Program to the community and develop strategies across programs to collaborate as a network. The CEP Council developed a written plan for training and monitoring and supported implementation of the training plan. CEP sites were provided with enrolled client lists.
  QI Program: The QI program is an evidence-based toolkit from prior studies that supported team leadership, case and care management, medication management, and CBT for Depression. The Case management manual supported depression screening and monitoring/tracking of outcomes; patient education and activation, care coordination, and behavioral activation and problem solving. The toolkit includes education on depression and a community health worker manual.
  CEP Council: The CEP Council was supported by a workbook de
Period: Overall Study
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Started | 606 (606 eligible clients enrolled and contacted by telephone for baseline or follow-up survey in RS arm) | 640 (640 eligible clients enrolled and contacted by telephone for baseline or follow-up survey in CEP arm)
Baseline | 492 | 489
6-Month Follow-Up | 380 | 379
12-Month Follow-Up | 364 | 369
3-Year Follow-up | 293 | 307
4-Year Follow-up (We attempted to contact 598 3-year participants who did not decline follow-up) | 143 | 140
Completed (Analytic sample comprises 1018 individuals who completed 1 or more surveys at baseline, 6 or 12 months with item level imputation for missing data and wave-level imputation for missing surveys.) | 504 (Clients in 44 programs with completed at least 1 data point at baseline, 6, or 12 mo FUP analyzed) | 514 (Clients in 46 programs with completed at least 1 data point at baseline, 6, or 12 mo FUP analyzed)
Not Completed | 102 | 126
Not completed — Withdrawal by Subject | 18 | 23
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 83 | 101

BASELINE CHARACTERISTICS:
Groups:
- Resources for Services RS: RS offers time-limited technical assistance to individual agencies and outreach from a community engagement specialty, to review components of the QI Program Intervention as implemented by the RS Expert Team.
  QI Program: The QI program is an evidence-based toolkit that supported team leadership, case and care management, medication management, and CBT for depression. The Case management manual supported depression screening and tracking of outcomes; patient education and activation, care coordination, and behavioral activation and problem solving. The toolkit includes education on depression and a community health worker manual. The expert team for RS consisted of 3 psychiatrists, a psychologist expert in CBT, a nurse care manager, a community engagement specialist, a QI expert, and staff support. The team offered 12 webinars to each community on components of collaborative care as well as site visits to primary care clinics on clinical assessment and medication management.
- Community Engagement and Planning CEP: CEP supports 4 months of planning for the CEP Council of representatives from assigned programs in biweekly 2-hr meetings to fit trainings in the QI Program to the community and develop strategies across programs to collaborate as a network. The CEP Council developed a written plan for training and monitoring and supported implementation of the training plan. CEP sites received enrolled client lists. The toolkit is the same as RS. The CEP Council was supported by a workbook developed by the overall CPIC Council that provided principles, approach, agendas, and resources for the multi-sector planning meetings. The CEP Councils met twice a month for 4-6 months to develop their plan and met monthly during implementation of trainings. The study Council supported CEP meetings. Community leaders co-led trainings with study experts to help assure sustainability. Each CEP council had $15K to defray costs of venues, materials, and consultations, while the study provided that for RS.
- Total: Total of all reporting groups
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP | Total
Number analyzed (Participants) | 504 | 514 | 1018
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (12.4) | 46.6 (13.2) | 45.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 309 | 595
  Male | 218 | 205 | 423
Race/Ethnicity, Customized [Number; unit: participants]
  Latino | 194 | 215 | 409
  African American | 239 | 249 | 488
  Non-Hispanic white | 45 | 41 | 86
  Other (Asian, Native American etc) | 26 | 9 | 35
Education [Number; unit: participants] — Note that the N's may differ slightly from published papers due to multiple imputation
  participants
    Less than high school education | 221 | 224 | 445
    High school or above | 283 | 290 | 573
Health Insurance Status [Number; unit: participants]
  No health insurance | 286 | 259 | 545
  Had health insurance | 218 | 255 | 473

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Poor Mental Health Quality of Life, MCS12≤ 40
Description: From the Short Form, 12-item quality of life measure, mental health-related quality of life is the primary client outcome. Poor mental health related quality of life is defined as MCS12≤ 40 (one standard deviation below population mean).
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 51.4 | 44.1
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a logistic regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 1,018 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority or Other; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.57 to 0.95]

2. Primary Outcome: Percent of Participants With PHQ-9 Score ≥ 10
Description: Patient Health Questionnaire 9-item version (PHQ-9) at least mild depression (score ≥ 10)
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 67.0 | 61.7
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.48 to 1.26]

3. Primary Outcome: Percent of Participants With Poor Mental Health Quality of Life, MCS12≤ 40
Description: as for outcome 1
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 50.5 | 44.8
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat analyses of repeated measures were developed including all participants with data at baseline, 6-month, or 12-month. Missing data were imputed. A generalized estimating equation (GEE) with a logit link function was used with adjustment for covariates; Test type: Superiority or Other; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.61 to 0.97]; In an analysis of change from baseline in likelihood of Poor Mental Health Quality of Life, CEP showed a significant advantage at 6 months, but not at 12 months

4. Primary Outcome: Percent of Participants With Poor Mental Health Quality of Life, MCS12≤ 40
Description: as for outcome 1
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 39.4 | 45.0
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using logistic regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 980 clients at 3 years to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.7 to 2.3]

5. Primary Outcome: Percent of Participants With PHQ-8 Score ≥ 10
Description: Patient Health Questionnaire 8-item version (PHQ-8) at least mild depression (score ≥ 10)
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 65.8 | 66.0
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a logistic regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 980 clients at 3 years to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.7]

6. Secondary Outcome: Percent of Participants With Mental Wellness
Description: Mental wellness is defined as at least a good bit of time in the prior 4 weeks on any of three items: feeling peaceful or calm, being a happy person, having energy
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 33.6 | 45.9
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.19 to 2.59]

7. Secondary Outcome: Percent of Participants Reported Organized Life
Description: A response of somewhat or definitely true to "my life is organized" versus unsure or somewhat false or definitely false
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 42.7 | 51.7
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.03 to 2.04]

8. Secondary Outcome: Percent of Participants With Physically Active
Description: Physically Active is defined as at least active to "How physically active you are?"
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 40.3 | 49.6
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.14 to 1.98]

9. Secondary Outcome: Percent of Participants With Homeless or ≥ 2 Risk Factors for Homelessness
Description: Defined as current homelessness or living in a shelter or having at least 2 risk factors (e.g., no place to stay for at least 2 nights or eviction from a primary residence, financial crisis, or food insecurity in the past 6 months)
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 39.8 | 29.7
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.38 to 0.96]

10. Secondary Outcome: Percent of Participants With Working for Pay
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 23.5 | 24.7
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.69 to 1.70]

11. Secondary Outcome: Percent of Participants With Any Missed Work Day in Last 30 Days, if Working
Time Frame: 6 months follow-up
Population: Population of individuals who are working
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 123 | 126
percentage of participants | 63.1 | 51.5
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Adjusted analyses used multiply imputed data (N= 249), weighted for eligible sample for enrollment; logistic regression model adjusted for baseline and covariates and accounted for the design effect of the cluster randomization; Test type: Superiority or Other; Odds Ratio (OR) = .59, 95% CI 2-sided [0.32 to 1.09]

12. Secondary Outcome: Percent of Participants With Hospitalization for Behavioral Health in the Past 6 Months
Description: self-reported services use in the past 6 months for overnight hospital stays for mental health or substance abuse
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 10.5 | 5.8
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.28 to 0.95]

13. Secondary Outcome: Percent of Participants With >=4 Hospital Nights for Behavioral Health in the Past 6 Months
Description: self-reported services use in the past 6 months with >=4 overnight hospital stays for any emotional, mental, alcohol, or drug problem, median cut point for baseline variable
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 5.8 | 2.1
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.14 to 0.88]

14. Secondary Outcome: Percent of Participants With >=2 Emergency Room Visits in the Past 6 Months
Description: self-reported services use in the past 6 months with >=2 emergency room visits in past 6 months, median cut point for baseline variable
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 512
percentage of participants | 28.3 | 24.5
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.52 to 1.25] — Median cut point for baseline variable

15. Secondary Outcome: Percent of Participants With Any MHS Outpatient Visit in the Past 6 Months
Description: self-reported mental health outpatient visit from mental health provider, including psychiatrists, psychologists, social workers, psychiatric nurses, or counselors in the past 6 months
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 53.9 | 53.6
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.69 to 1.41]

16. Secondary Outcome: Percent of Participants With Any PCP Visit With Depression Service in the Past 6 Months
Description: self-reported services use in the past 6 months with any primary care visit for depression
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 29.2 | 29.4
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using logistic regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 1,018 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority or Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.70 to 1.46]

17. Secondary Outcome: Percent of Participants With >= 2 PCP Visits With Depression Services, if Any
Time Frame: 6 months follow-up
Population: Individuals who reported any PCP visit in past 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 145 | 153
percentage of participants | 61.9 | 79.8
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Adjusted analyses used multiply imputed data (N=298), weighted for eligible sample for enrollment; logistic regression model adjusted for baseline and covariates and accounted for the design effect of the cluster randomization; Test type: Superiority or Other; p < .01, Regression, Logistic; Odds Ratio (OR) = 2.63, 95% CI 2-sided [1.40 to 4.94]

18. Secondary Outcome: Percent of Participants With Faith-based Program Participation in the Past 6 Months
Description: Went to any religious or spiritual places such as a church, mosque, temple, or synagogue in the past 6 months
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 59.5 | 57.1
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a generalized estimating equation logistic regression model adjusted for covariates, accounted for the design effect of the cluster randomization. We weighted data for 1,018 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority or Other; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.66 to 1.21]

19. Secondary Outcome: Percent of Participants With Any Use of Park and Recreation or Community Centers in the Past 6 Months
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 41.1 | 39.4
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.61 to 1.40]

20. Secondary Outcome: Percent of Participants With Use of an Antidepressant Medication for 2 Months or More in the Past 6 Months
Time Frame: 6 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
percentage of participants | 39.2 | 31.5
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.34 to 1.25]

21. Secondary Outcome: Medication Visits Among MHS Users in the Past 6 Months
Time Frame: 6 months follow-up
Population: Individuals who reported any mental health specialty outpatient visit in past 6 months
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 276 | 277
visits | 10.9 [6.2 to 15.5] | 5.3 [4.1 to 6.6]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Adjusted analyses used multiply imputed data (N=553), weighted for eligible sample for enrollment; Poisson regression model adjusted for baseline and covariates and accounted for the design effect of the cluster randomization; Test type: Superiority or Other; Rate Ratio (RR) = 0.49, 95% CI 2-sided [0.30 to 0.82]

22. Secondary Outcome: Faith-based Visits With Depression Service if Faith Participation in the Past 6 Months
Description: For this sector, depression/mental health service is defined by client report of having assessment, counseling, education, medication discussion or referral for depression or emotional or mental health problems.
Time Frame: 6 months follow-up
Population: Individuals who reported any faith based participation in past 6 months
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 299 | 289
visits | 0.7 [0.3 to 1.0] | 1.9 [0.9 to 2.9]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Adjusted analyses used multiply imputed data (N=588), weighted for eligible sample for enrollment; Poisson regression model adjusted for baseline status of the dependent variable and covariates and accounted for the design effect of the cluster randomization; Test type: Superiority; Rate Ratio (RR) = 2.84, 95% CI 2-sided [1.39 to 5.80]

23. Secondary Outcome: Park or Community Center Visits With Depression Service if Went to Park or Community Center in Past 6 Months
Description: as for outcome 22
Time Frame: 6 months follow-up
Population: Individuals who reported any park or community center visit in past 6 months
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 210 | 199
visits | 0.3 [0.0 to 0.5] | 1.6 [0.2 to 3.1]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Adjusted analyses used multiply imputed data (N=410), weighted for eligible sample for enrollment; Poisson regression model adjusted for baseline and covariates and accounted for the design effect of the cluster randomization; Test type: Superiority or Other; Rate Ratio (RR) = 6.20, 95% CI 2-sided [1.5 to 24.9]

24. Secondary Outcome: Total Mental Health Related Outpatient Visits in the Past 6 Months
Description: Total outpatient visits for depression, mental health or substance abuse from emergency rooms, primary care or public health, mental health, substance abuse, or social-community services sectors in the past 6 months
Time Frame: 6 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 504 | 514
visits | 22.9 [14.8 to 30.9] | 21.9 [16.3 to 27.4]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a Poisson regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 1,018 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority or Other; Rate Ratio (RR) = 0.96, 95% CI 2-sided [0.59 to 1.57]

25. Secondary Outcome: Percent of Participants With Hospitalization for Behavioral Health in the Past 6 Months
Description: self-reported services use in the past 6 months for overnight hospital stays for mental health or substance abuse
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 5.0 | 4.3
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 0.70, 95% CI 2-sided [.40 to 1.22] — When analyzed as change from baseline, CEP showed significant reductions in likelihood of behavioral health hospitalizations at 6 months (P < 0.01) and 12 months (P < 0.01)

26. Secondary Outcome: Percent of Participants With Any MHS Outpatient Visit in the Past 6 Months
Description: as for outcome 15
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 44.5 | 42.6
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.05, 95% CI 2-sided [.66 to 1.66]

27. Secondary Outcome: Percent of Participants With Any PCP Visit With Depression Service in the Past 6 Months
Description: self-reported services use in the past 6 months with any primary care visit for depression
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 25.1 | 28.4
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.74 to 1.42]

28. Secondary Outcome: Percent of Participants With Faith-based Program Participation in the Past 6 Months
Description: Went to any religious or spiritual places such as a church, mosque, temple, or synagogue in the past 6 months
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 57.0 | 53.9
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = .79, 95% CI 2-sided [.60 to 1.05]

29. Secondary Outcome: Percent of Participants With Any Use of Park and Recreation or Community Centers in the Past 6 Months
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 34.5 | 36.6
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = .97, 95% CI 2-sided [0.72 to 1.32]

30. Secondary Outcome: Percent of Participants With Use of an Antidepressant Medication for 2 Months or More in the Past 6 Months
Time Frame: 12 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
percentage of participants | 34.0 | 28.7
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; Odds Ratio (OR) = .87, 95% CI 2-sided [0.55 to 1.39]

31. Secondary Outcome: Total Mental Health Related Outpatient Visits in the Past 6 Months
Description: as for outcome 24
Time Frame: 12 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 501 | 512
visits | 18.7 [13.6 to 23.8] | 17.0 [12.0 to 22.1]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat analyses of repeated measures were developed including all participants with data at baseline, 6-month, or 12-month. Missing data were imputed. A generalized estimating equation (GEE) with a log link function was used with adjustment for covariates; Test type: Superiority or Other; Rate Ratio (RR) = .91, 95% CI 2-sided [0.65 to 1.29]

32. Secondary Outcome: PCS-12 Scores on 12-Item Physical Health Summary Measure, Comparison Between CEP and RS Groups
Description: 12-item physical composite score (PCS-12). Possible scores on range from 0 to 100, with higher scores indicating better physical health
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
units on a scale | 38.7 [37.9 to 39.5] | 39.9 [39.2 to 40.6]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a linear regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 980 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.2 to 2.0]

33. Secondary Outcome: Nights Hospitalized for Behavioral Health Reason in the Past 6 Months
Description: self-reported number of overnight hospital stays for any emotional, mental, alcohol, or drug problem in past 6 months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: nights
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
nights | 1.2 [0.3 to 4.6] | 0.2 [0.1 to 0.4]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a Poisson regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 980 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority; Rate Ratio (RR) = 0.2, 95% CI 2-sided [0.1 to 0.8]

34. Secondary Outcome: N of Emergency Room or Urgent Care Visits in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
visits | 1.5 [1.0 to 2.2] | 1.9 [0.7 to 4.9]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.2, 95% CI 2-sided [0.4 to 3.7]

35. Secondary Outcome: N of Visits to Primary Care in Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
visits | 3.9 [2.7 to 5.4] | 4.1 [3.5 to 4.9]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.1, 95% CI 2-sided [0.8 to 1.5]

36. Secondary Outcome: N of Outpatient Visits to Primary Care for Depression Services in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
visits | 1.1 [0.6 to 2.1] | 1.1 [0.8 to 1.5]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.0, 95% CI 2-sided [0.5 to 2.1]

37. Secondary Outcome: N of Outpatient Mental Health Visits in Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
visits | 5.5 [3.7 to 8.0] | 5.6 [3.2 to 9.8]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.0, 95% CI 2-sided [0.7 to 1.6]

38. Secondary Outcome: N of Outpatient Visits to a Substance Abuse Treatment Agency or Self Help Group in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
visits | 11.1 [4.7 to 24.5] | 12.3 [5.6 to 25.8]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.1, 95% CI 2-sided [0.3 to 4.0]

39. Secondary Outcome: N of Social Services for Depression Visits in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: visits
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
visits | 0.6 [0.3 to 1.2] | 0.6 [0.4 to 0.9]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.1, 95% CI 2-sided [0.4 to 2.7]

40. Secondary Outcome: Number of Calls to Hotline for Substance Use or Mental Health Problem in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: calls
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
calls | 0.2 [0.1 to 0.6] | 0.3 [0.1 to 1.1]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 1.4, 95% CI 2-sided [0.2 to 8.6]

41. Secondary Outcome: N of Days on Which a Self-help Visit for Mental Health Was Made in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
days | 6.3 [4.1 to 9.6] | 5.6 [3.4 to 9.1]
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; Rate Ratio (RR) = 0.9, 95% CI 2-sided [0.4 to 1.8]

42. Secondary Outcome: Percent of Participants With Any Faith-based Services for Depression in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 9.4 | 15.2
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a logistic regression model adjusted for baseline and covariates, and accounted for the design effect of the cluster randomization. We weighted data for 980 clients to characteristics of the eligible sample, with item-level imputation for missing data and wave-level imputation for missing surveys. Weights account for non-enrollment among eligible clients and attrition; Test type: Superiority; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.2 to 2.6]

43. Secondary Outcome: Percent of Participants With Use of Any Antidepressant in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 28.7 | 26.9
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.5 to 1.5]

44. Secondary Outcome: Percent of Participants With Use of Any Mood Stabilizer in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 2.5 | 6.4
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 2.9, 95% CI 2-sided [1.0 to 8.3]

45. Secondary Outcome: Percent of Participants With Use of Any Antipsychotic in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 21.7 | 23.4
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.7 to 1.7]

46. Secondary Outcome: Percent of Participants With Any Visit in Health Care Sector in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 84.2 | 84.3
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.5 to 2.0]

47. Secondary Outcome: Percent of Participants With Any Community-sector Visit for Depression in the Past 6 Months
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 28.3 | 35.6
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.4, 95% CI 2-sided [1.0 to 2.0]

48. Secondary Outcome: Percent of Participants With Any Depression Treatment in the Past 6 Months
Description: Antidepressant use for at least two months or at least four outpatient visits to mental health or primary care setting for depression services
Time Frame: 36 months follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 483 | 497
percentage of participants | 43.2 | 43.5
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 42, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.6 to 1.7]

49. Secondary Outcome: Survival Analysis for Time to the First Clinical Remission
Description: clinical remission: Patient Health Questionnaire, PHQ-8 score <10. Cox Proportional Hazard model was used to examine the impact of the intervention on speed of clinical remission over the 3 years follow-up period, defined as the first assessment with clinical remission (PHQ-8<10).
Time Frame: from baseline to 3 years
Population: Sample does not include persons in clinical remission at baseline
Measure: Mean (Standard Deviation); unit: months to remission
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 491 | 504
months to remission | 21.14 (13.98) | 20.05 (14.14)
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a Cox proportional-hazards model adjusted for baseline covariates. Data were multiply imputed and weighted for eligible sample for enrollment, accounted for the design effect of the cluster randomization; Test type: Superiority; p > .05, Regression, Cox; Cox Proportional Hazard = 1.12, 95% CI 2-sided [0.83 to 1.50]

50. Secondary Outcome: Survival Analysis for Time to the First Community-Defined Remission
Description: Community-Defined Remission: PHQ-8<10 or MCS-12>40 or any mental wellness. Cox Proportional Hazard model was used to examine the impact of the intervention on speed of community-defined remission over the 3 years follow-up period, defined as the first assessment with community-defined (PHQ-8<10 or MCS-12>40 or any mental wellness)
Time Frame: from baseline to 3 years
Population: Sample does not include persons in community-defined remission at baseline
Measure: Mean (Standard Deviation); unit: months to remission
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 203 | 205
months to remission | 14.05 (11.97) | 12.14 (10.93)
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p > 0.05, Regression, Cox; Cox Proportional Hazard = 1.23, 95% CI 2-sided [0.99 to 1.52]

51. Secondary Outcome: Percent of Participants With Clinical Remission
Description: Clinical remission defined as Patient Health Questionnaire-2 (PHQ-2) score < 3.
Time Frame: 4 years follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 143 | 140
percentage of participants | 39.7 | 51.7
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; Intent-to-treat, comparative-effectiveness analyses with intervention status as the independent variable, using a logistic regression model adjusted for baseline covariates. Data were multiply imputed and weighted for eligible sample for enrollment, accounted for the design effect of the cluster randomization; Test type: Superiority; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.00 to 2.99]

52. Secondary Outcome: Percent of Participants With Community-Defined Remission
Description: Community-Defined Remission defined as PHQ-2<3, MCS-12>40, or mental wellness
Time Frame: 4 years follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
Number analyzed (Participants) | 143 | 140
percentage of participants | 69.0 | 84.2
Statistical Analysis 1: Comparison: Resources for Services RS vs Community Engagement and Planning CEP; [analysis description as in outcome 51, analysis 1]; Test type: Superiority; Odds Ratio (OR) = 2.62, 95% CI 2-sided [1.24 to 5.54]

ADVERSE EVENTS:
Time Frame: Mortality data obtained from back up contact person identified by participants in prior survey periods. The suicidal ideation within the last two weeks data was collected over the 12 months study duration.
Description: Screening for suicidal ideation in the baseline utilized the Mini-International Neuropsychiatric Interview (MINI) item: "Over the past two weeks, when you felt depressed or uninterested, did you repeatedly consider hurting yourself, feel suicidal, or wish that you were dead? Did you attempt suicide or plan a suicide? At 6 and 12 months, screening utilized the item 9 of the Patient Health Questionnaire with a follow-up question: "Are these thoughts bothering you now?" if responding affirmatively.
Arm/Group | Resources for Services RS | Community Engagement and Planning CEP
All-Cause Mortality (participants affected / at risk) | 4/606 | 4/640
Serious Adverse Events (participants affected / at risk) | 0/606 | 0/640
Other Adverse Events (participants affected / at risk) | 126/606 | 126/640
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resources for Services RS (N=606) | Community Engagement and Planning CEP (N=640)
Suicidality Screening Tool (MINI) at baseline (Psychiatric disorders) | 76 | 67 — Over the past two weeks, when you felt depressed or uninterested, did you repeatedly consider hurting yourself, feel suicidal, or wish that you were dead? Did you attempt suicide or plan a suicide?
Suicidal ideation on the 9 item of PHQ-9 at 6 months (Psychiatric disorders) | 53 | 46 — the 9 item of Patient Health Questionnaire (PHQ-9): In the past two weeks, have you been bothered by thoughts that you would be better off dead or of hurting yourself in some way?
Suicidal ideation on the 9 item of PHQ-9 with positive follow-up at 6 months (Psychiatric disorders) | 13 | 16 — a participant responding affirmatively to the 9 item of PHQ-9 answered "yes" to the follow-up question: "Are these thoughts bothering you now?"
Suicidal ideation on the 9 item of PHQ-9 at 12 months (Psychiatric disorders) | 72 | 74 — the 9 item of Patient Health Questionnaire (PHQ-9): In the past two weeks, have you been bothered by thoughts that you would be better off dead or of hurting yourself in some way?
Suicidal ideation on the 9 item of PHQ-9 with positive follow-up at 12 months (Psychiatric disorders) | 23 | 21 — a participant responding affirmatively to the 9 item of PHQ-9 answered "yes" to the follow-up question: "Are these thoughts bothering you now?"

LIMITATIONS AND CAVEATS:
Communities had history of using CPPR for depression. Response rates moderate for agencies, high for programs. Convenience samples of sites. Client retention rates lower than other QI studies. Outcomes rely on client self-report at 6-month follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT01699789/Prot_SAP_ICF_000.pdf